CLINICAL TRIAL: NCT02022384
Title: Immunophenotyping From Blood From Patients With Glioblastoma and Anaplastic Astrocytoma Before and During Chemoradiation as Well as During Adjuvant Chemotherapy
Brief Title: Immunophenotyping From Blood of Patients With Malignant Gliomas
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: IMMO-GLIO 01
Record Dates: First submitted 2013-12-13; First posted 2013-12-27 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Anaplastic Astrocytoma; Glioblastoma Multiforme
Keywords: Malignant glioma; Anaplastic astrocytoma; Glioblastoma multiforme; Immune; Immunophenotyping; Immune cells; activation state; Quality of live; translational research
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Glioma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study patients: Blood sample and life quality questionnaires
  Interventions: Other: Blood sample and life quality questionnaires

INTERVENTIONS:
Other: Blood sample and life quality questionnaires — Blood will be drawn at distinct time points during and after radio(chemo)therapy

SUMMARY:
In this explorative study immunological changes during tumor therapy will be analyzed in patients with malignant glioma. Immunophenotyping before and during therapy is used as analysis method. Thereby immune cells are quantitatively and qualitatively detected from patient's blood at continuous time points. Additionally relevant mediators like cytokines, danger signals and chemokines are analyzed by other methods. Obtained results may give information about the effects of therapy on immunological processes and immune cells and may help to find immunological based predictive or prognostic tumor markers and to define time points for including additional immune therapy in the future.

DETAILED DESCRIPTION:
Patients with malignant glioma generally have a bad prognosis. To improve patients' situation new therapy options as well as new possibilities to determine prognosis and prediction more precisely are needed. One approach is the targeted activation of the immune system to recognize and eliminate tumor cells. Due to cerebral tumors the brain is no immune privileged organ anymore, so that immune cells may pass the haemato-encephalic barrier to attack tumor cells. This study aims to offer valuable clues about how the immune system is influenced by standard therapies (radiotherapy and chemotherapy). Just with the background knowledge of immune mechanisms and influencing factors by tumor therapy, an effective anti-tumor response can systematically be induced by modulating immune therapy. To analyze immunological changes, immunophenotyping by flow cytometry is performed with blood from patients with malignant gliomas during their therapy concluding chemoradiation and chemotherapy alone. Count, class and activation status of immune cells are detected by flow cytometry. Together with additional analysis methods, information about immunological mediators like cytokines, chemokines and danger signals can be received. For these purposes serum and plasma are generated from blood samples and stored for prospective questions. The explorative determined results may also help to discover new, immunological based, prognostic or predictive tumor markers.

ELIGIBILITY:
Inclusion Criteria:

* patients with glioblastoma or anaplastic astrocytoma
* legal age
* planned chemoradiation and adjuvant chemotherapy (according to Stupp et. al.)

Exclusion Criteria:

* Fertile patients who refuse effective contraception during study treatment
* persistent drug and/or alcohol abuse
* patients not able or willing to behave according to study protocol
* patients in care
* patients that are not able to speak German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with primary diagnosed glioblastoma multiforme or anaplastic astrocytoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
immunological state of patients comprising number, type and activation state of immune cells, cytokines and danger signals from peripheral blood | patients will be followed for the duration of therapy and follow-up until recurrence, an expected average of 6 months
  Time points for blood sample collections:
  Before start of chemoradiation (RCT). In 3th week of RCT. At last day of RCT. At the beginning of chemotherapy (CT) (about 4 weeks after RCT). During CT each three to four weeks. At follow-up visits each one to three months. During recurrence therapy.

SECONDARY OUTCOMES:
Acquisition of toxicities according to Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | patients will be followed for the duration of therapy and follow-up until recurrence, an expected average of 6 months
documentation of medication | patients will be followed for the duration of therapy and follow-up until recurrence, an expected average of 6 months
Acquisition of changes in imaging | patients will be followed for the duration of therapy and follow-up until recurrence, an expected average of 6 months
Acquisition of life quality according to quality of life questionnaire (QLQ) (EORTC QLQ -BN20) | patients will be followed for the duration of therapy and follow-up until recurrence, an expected average of 6 months
correlation of immunological parameters with clinical data | patients will be followed for the duration of therapy and follow-up until recurrence, an expected average of 6 months
  Correlation with results of immunophenotyping, possibly definition of medically relevant markers
overall survival | patients will be followed for the duration of therapy and follow-up until recurrence, an expected average of 6 months
progression free survival | patients will be followed for the duration of therapy and follow-up until recurrence, an expected average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, Prof., Principal Investigator — Department of Radiation Oncology, Universitätsklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg; Udo S Gaipl, Prof., Principal Investigator — Department of Radiation Oncology, Universitätsklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- Departement of Radiation Oncology, Universitätsklinikum Erlangen, Friedrich-Alexander-Universität erlangen-Nürnberg, Erlangen, BAY, Germany

REFERENCES:
- [Derived] Ruhle PF, Goerig N, Wunderlich R, Fietkau R, Gaipl US, Strnad A, Frey B. Modulations in the Peripheral Immune System of Glioblastoma Patient Is Connected to Therapy and Tumor Progression-A Case Report from the IMMO-GLIO-01 Trial. Front Neurol. 2017 Jun 23;8:296. doi: 10.3389/fneur.2017.00296. eCollection 2017. PMID 28690586